CLINICAL TRIAL: NCT05859932
Title: A Look at the Patterns in Clinical Research Participation Among Patients With Hairy Cell Leukemia
Brief Title: Assessing Medical Trial Experiences of Hairy Cell Leukemia Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 81405664
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Hairy Cell Leukemia
Keywords: hairy cell leukemia
MeSH Terms: conditions — Leukemia, Hairy Cell

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The percentages of participants in clinical studies haven't always been perfectly representative of a particular group.

This research examines the variables that affect a patient's choice to enroll in, discontinue participation in, or resume participation in a clinical trial for hairy cell leukemia.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of hairy cell leukemia studies.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* Ability to understand and the willingness to sign a written informed consent document.
* Willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.

Exclusion Criteria:

* Is pregnant, breastfeeding or expecting to conceive within the projected duration of the study
* Any mental or medical condition that prevents the patient from giving informed consent or participating in the trial
* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are actively considering involvement in an observational hairy cell leukemia clinical trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a hairy cell leukemia clinical study. | 3 months
Number of hairy cell leukemia study participants who remain in clinical trial until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chihara D, Arons E, Stetler-Stevenson M, Yuan CM, Wang HW, Zhou H, Raffeld M, Xi L, Steinberg SM, Feurtado J, James L, Wilson W, Braylan RC, Calvo KR, Maric I, Dulau-Florea A, Kreitman RJ. Randomized Phase II Study of First-Line Cladribine With Concurrent or Delayed Rituximab in Patients With Hairy Cell Leukemia. J Clin Oncol. 2020 May 10;38(14):1527-1538. doi: 10.1200/JCO.19.02250. Epub 2020 Feb 28. PMID 32109194
- [Background] Maitre E, Paillassa J, Troussard X. Novel targeted treatments in hairy cell leukemia and other hairy cell-like disorders. Front Oncol. 2022 Dec 22;12:1068981. doi: 10.3389/fonc.2022.1068981. eCollection 2022. PMID 36620555
- [Background] Kreitman RJ. Hairy cell leukemia: present and future directions. Leuk Lymphoma. 2019 Dec;60(12):2869-2879. doi: 10.1080/10428194.2019.1608536. Epub 2019 May 9. PMID 31068044

DOCUMENTS (1):
  • Informed Consent Form (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/32/NCT05859932/ICF_000.pdf